CLINICAL TRIAL: NCT07159672
Title: Prospective Cohort Study of Nutritional, Metabolic, Molecular, and Volumetric Assessment of the Remnant Pancreas in Patients With Periampullary Malignancies Undergoing Pancreaticoduodenectomy
Brief Title: Cohort Study on Nutritional, Metabolic, and Volumetric Assessment After Pancreaticoduodenectomy
Status: Completed | Type: Observational
Sponsor: Marco Aurélio Ribeiro, PhD (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Sponsor-Investigator, Marco Aurélio Ribeiro, PhD, Principal Investigator, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Other Study IDs: 64695422.6.0000.5440; 88887.827259/2023-00 (Other Grant/Funding Number: CAPES); 141784/2025-3 (Other Grant/Funding Number: CNPq); Finance Code 001 (Other Grant/Funding Number: CAPES); 63993522.3.0000.5440 (Registry Identifier: Certificado de Apresentação para Apreciação Ética (CAAE)); 64695422.6.0000.5440 (Registry Identifier: Certificado de Apresentação para Apreciação Ética (CAAE))
Record Dates: First submitted 2025-08-22; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Periampullary Neoplasms; Pancreatic Cancer; Pancreaticoduodenectomy
Keywords: Nutritional Assessment; Resting Energy Expenditure; Bioimpedance Analysis; Molecular Biomarkers; Oxidative Stress; Proteomics; Lipidomics; Pancreatic Volume; 3D Imaging / 3D Slicer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pancreaticoduodenectomy Group: Patients aged 18-80 years with periampullary malignant neoplasms undergoing pancreaticoduodenectomy (classic Whipple or pylorus-preserving). This group will be followed prospectively for nutritional, metabolic, molecular, and volumetric assessments at baseline (preoperative), 3 months, and 6 months after hospital discharge.
  Interventions: Procedure: Pancreaticoduodenectomy
- Control Group: Age- and sex-matched individuals without malignant gastrointestinal disease, selected among those undergoing routine upper gastrointestinal endoscopy with normal or nonspecific findings. This group will undergo a single-time evaluation for nutritional, metabolic, molecular, and imaging parameters.

INTERVENTIONS:
Procedure: Pancreaticoduodenectomy — Pancreaticoduodenectomy (classic Whipple or pylorus-preserving) performed as part of standard clinical care for patients with periampullary malignant neoplasms. This procedure is not assigned by the study protocol, but is the exposure of interest. The study observes nutritional, metabolic, molecular, and imaging outcomes at baseline (preoperative), and at 3 and 6 months after hospital discharge.
  Other Names: Whipple procedure; Pylorus-preserving pancreaticoduodenectomy
  Groups: Pancreaticoduodenectomy Group

SUMMARY:
Periampullary malignant neoplasms are among the most lethal gastrointestinal tumors. They are usually diagnosed at advanced stages and require complex surgical treatment. Pancreaticoduodenectomy, the standard procedure for resectable cases, significantly impacts nutritional status, pancreatic function, and the structural integrity of the remaining pancreas. However, there are still significant knowledge gaps regarding the volumetric and molecular changes that occur postoperatively and how these changes interact with body composition, resting energy expenditure, and biochemical markers.

This prospective, controlled, cohort study aims to integrate clinical, nutritional, metabolic, molecular, and imaging data to investigate changes in the remnant pancreas and their associations with postoperative outcomes. The study is expected to provide novel insights to support personalized, evidence-based nutritional and metabolic care for patients undergoing pancreaticoduodenectomy.

DETAILED DESCRIPTION:
Periampullary malignant neoplasms are lethal gastrointestinal tumors that are often diagnosed at advanced stages and require complex surgical intervention. Pancreaticoduodenectomy, the gold standard for resectable disease, has profound effects on nutritional status, exocrine pancreatic function, and the structural integrity of the remaining pancreas. Despite recent advances, significant gaps remain in our understanding of the volumetric and molecular alterations that occur postoperatively and how these alterations interact with body composition, resting energy expenditure, and biochemical markers.

This is a prospective, longitudinal, controlled, clinical-translational cohort study. Data on clinical, nutritional, biochemical, and plasma parameters will be collected at three time points for the experimental group (preoperatively and 3 and 6 months after hospital discharge) and one time point for the control group. Plasma samples will be stored at -80 °C and analyzed using validated techniques, including multiplex assays, spectrophotometry, ELISA, and tandem mass spectrometry (LC-MS/MS) to detect inflammatory biomarkers (IL-1β, , IL-6, TNF-α, and MCP-1; oxidative markers (MDA, GSH, TAC, and FRAP); proteomic targets (HSP70, fibronectin, and laminin); and lipidomic profiles (ceramides, sphingolipids, and cardiolipins). Abdominal imaging (CT and/or MRI) will be processed using 3D Slicer software to estimate the volume of the remnant pancreas via three-dimensional segmentation.

Statistical analyses will be conducted in RStudio. We will apply mixed linear models (MLM and MLMG), incorporating fixed and random effects to account for intra- and inter-individual variability. Missing not-at-random data will be addressed using multiple imputation by chained equations (MICE), and pooled estimates will be calculated according to Rubin's rules. We will set statistical significance at p < 0.05 with Holm-Bonferroni correction for multiple comparisons.

This integrative approach ensures methodological rigor, bias control, and robust inference. It has the potential to guide personalized, evidence-based nutritional strategies in the context of pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 80 years;
* Histologically or radiologically confirmed diagnosis of resectable periampullary malignant neoplasms (e.g., pancreatic head adenocarcinoma, ampullary carcinoma, distal cholangiocarcinoma, duodenal adenocarcinoma);
* Candidates for elective pancreaticoduodenectomy (either classic Whipple or pylorus-preserving technique), performed by the institutional surgical team following standardized protocols;
* ECOG Performance Status ≤2;
* Adequate cardiopulmonary function to undergo major surgery, as assessed preoperatively;
* Ability and willingness to provide written informed consent.

Exclusion Criteria:

* Previous pancreatic surgery;
* Pancreaticoduodenectomy performed outside the study institution;
* Evidence of unresectable disease, distant metastases, or local tumor recurrence at baseline imaging or intraoperative assessment;
* Active inflammatory or autoimmune diseases (e.g., rheumatoid arthritis, lupus, inflammatory bowel disease);
* Active malignancy other than periampullary cancer, or history of non-pancreatic cancer within the past 5 years;
* Use of systemic immunosuppressive therapy (e.g., corticosteroids >10 mg/day prednisone equivalent, chemotherapy, biologics);
* Diagnosed malabsorption syndromes unrelated to pancreatic disease;
* Severe hepatic dysfunction or severe renal impairment (eGFR <30 mL/min/1.73m²);
* Pregnancy or breastfeeding;
* Refusal or inability to attend scheduled follow-up visits within 6 months;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 44 individuals.
  The experimental group will include 24 adults aged 18-80 years with histologically or radiologically confirmed resectable periampullary malignant neoplasms (e.g., pancreatic head adenocarcinoma, ampullary carcinoma, distal cholangiocarcinoma, duodenal adenocarcinoma), undergoing pancreaticoduodenectomy (classic Whipple or pylorus-preserving), performed by the same institutional surgical team with standardized techniques (end-to-side duct-to-mucosa pancreaticojejunostomy). Participants will be evaluated at baseline (preoperative), 3 months, and 6 months post-discharge.
  The control group will include 20 age- and sex-matched individuals without gastrointestinal malignancy, selected among patients undergoing routine upper GI endoscopy with normal or nonspecific findings. Control subjects will be assessed once. All procedures will follow standardized clinical, nutritional, and laboratory protocols.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Resting Energy Expenditure (REE) in kcal/day | Day 0 (preoperative), 3 months post-discharge, and 6 months post-discharge
  Resting energy expenditure will be measured using indirect calorimetry (Quark RMR®) following standardized protocols. Results will be expressed in kcal/day, and normalized to body weight and fat-free mass. Results will be compared with predictive equations (Harris-Benedict, Mifflin-St Jeor, FAO/WHO).

SECONDARY OUTCOMES:
Fat-Free Mass (kg) measured by multifrequency bioimpedance analysis | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Fat-free mass will be assessed using multifrequency bioimpedance (SECA mBCA 525®). Values will be reported in kilograms and normalized by body surface area.
Fat Mass (kg) measured by multifrequency bioimpedance analysis | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Fat mass will be measured using SECA mBCA 525® bioimpedance. Results will be expressed in kilograms and monitored across study visits.
Hydration Status (%) assessed by bioimpedance analysis | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Percentage of total body water will be determined by SECA mBCA 525® device using multifrequency bioimpedance.
Phase Angle (°) assessed by bioimpedance analys | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Phase angle will be derived from resistance and reactance using multifrequency BIA with SECA mBCA 525®, as a proxy of cell membrane integrity.
Total Serum Protein (g/dL) | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Measured using colorimetric assay with spectrophotometric reading at 540 nm. Reference range: 6.0-8.3 g/dL.
Serum Albumin (g/dL) | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Quantified using specific colorimetric method with reading at 625 nm. Normal range: 3.5-5.0 g/dL.
Serum C-Reactive Protein - CRP (mg/L) | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Systemic inflammation marker measured via immunoturbidimetric assay with latex particles. Reference value: <3 mg/L.
Fasting Glucose (mg/dL) | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Measured by enzymatic colorimetric method. Reference range: 70-99 mg/dL.
Hemoglobin (g/dL) | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Determined by automated hematology analyzer (ABX Pentra DX120), using impedance, photometry, and fluorescence. Reference: 13-17.5 g/dL (men), 12-15.5 g/dL (women).
Absolute Lymphocyte Count (×10³/mm³) | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Analyzed using automated hematology analyzer. Normal range: 1.0-4.0 ×10³/mm³.
Serum Iron (µg/dL) | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Determined by direct colorimetric method. Normal range: 65-175 µg/dL (men), 50-170 µg/dL (women).
Serum Ferritin (ng/mL) | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Measured by chemiluminescence (Immulite 2000). Normal: 30-300 ng/mL (men), 15-150 ng/mL (women).
Latent Iron-Binding Capacity - LIBC (µg/dL) | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Assessed via direct colorimetric method. Reference: 240-450 µg/dL.
Serum Transferrin (mg/dL) | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Calculated using Vannucchi et al. (1996): Transferrin = ((LIBC + Iron) × 0.8) - 43. Reference: 200-360 mg/dL.
Transferrin Saturation (%) | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Calculated by serum iron / LIBC ratio. Normal range: 20-50%.
Serum Urea (mg/dL) | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Measured using kinetic method and spectrophotometric reading at 340 nm. Reference: 10-40 mg/dL.
Serum Creatinine (mg/dL) | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Quantified by kinetic method with reading at 500 nm. Reference: 0.7-1.3 mg/dL (men), 0.6-1.1 mg/dL (women).
AST (U/L) | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Aspartate aminotransferase assessed via optimized UV method. Normal range: 10-40 U/L.
ALT (U/L) | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Alanine aminotransferase determined by UV method at 340 nm. Reference: 7-56 U/L.
Serum Folate - Vitamin B9 (ng/mL) | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Measured by chemiluminescence (Immulite 2000). Reference: 3.0-17.0 ng/mL.
Serum Vitamin B12 (pg/mL) | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Cobalamin levels determined by chemiluminescence. Normal range: 200-900 pg/mL.
Vitamin A - Retinol (µg/dL) | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Determined by HPLC. Reference: 30-80 µg/dL.
Vitamin E - Alpha-tocopherol (mg/dL) | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Assessed by HPLC. Normal range: 0.5-2.0 mg/dL.
Plasma Copper (µg/dL) | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Measured by atomic absorption spectroscopy at 327.4 nm. Reference: 70-140 µg/dL (men), 80-155 µg/dL (women).
Plasma Zinc (µg/dL) | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Determined via atomic absorption spectroscopy at 213.9 nm. Reference: 60-120 µg/dL.
Sudan III Stool Test (qualitative) | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Microscopic evaluation of Sudan III-stained stool samples for detection of steatorrhea. Reported as positive or negative.
Interleukin 1 beta (IL-1β), pg/mL | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Plasma concentrations will be quantified using a multiplex immunoassay with magnetic beads (MagPix®, Luminex Corporation), following manufacturer's specifications.
Interleukin 4 (IL-4), pg/mL | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Quantified via bead-based multiplex fluorescence assay using the MagPix® system (Luminex®), allowing simultaneous detection of multiple cytokines.
Interleukin 6 (IL-6), pg/mL | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Measured by high-sensitivity magnetic bead-based immunoassay (Luminex® MagPix®), using standard calibration curves.
Interleukin 8 (IL-8), pg/mL | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Determined using multiplex fluorescence-based immunoassay with magnetic bead differentiation and spectral laser detection.
Interleukin 10 (IL-10), pg/mL | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Plasma levels will be assessed using a validated multiplex Luminex® panel, enabling parallel cytokine detection.
Tumor Necrosis Factor Alpha (TNF-α), pg/mL | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Measured by multiplex immunoassay with magnetic beads on the Luminex® platform; assay sensitivity <1 pg/mL.
Interferon Gamma (INF-γ), pg/mL | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Quantified using bead-based multiplex immunoassay with MagPix® system and fluorophore-labeled secondary antibodies.
Vascular Endothelial Growth Factor (VEGF), pg/mL | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Determined by multiplex immunoassay using magnetic beads, with detection by Luminex® MagPix® laser-based fluorescence reader.
Monocyte Chemoattractant Protein 1 (MCP-1), pg/mL | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Assessed using a Luminex®-based multiplex immunoassay with internal controls and duplicate sampling.
Free Plasma Amino Acids (HPLC), nmol/mL | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Quantified by high-performance liquid chromatography (HPLC) with pre-column derivatization using o-phthaldialdehyde (OPA) and fluorescence detection (excitation: 340 nm; emission: 450 nm).
Malondialdehyde (MDA), nmol/mL | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Measured by the thiobarbituric acid reactive substances (TBARS) assay, with spectrophotometric reading at 532 nm.
Reduced Glutathione (GSH), µmol/L | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Quantified by spectrophotometric method using DTNB (5,5'-dithiobis-(2-nitrobenzoic acid)), with absorbance measured at 412 nm.
Total Hydroperoxides (FOX), µmol/L | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Measured using the Ferrous Oxidation-Xylenol Orange (FOX) method with absorbance at 560 nm.
Total Antioxidant Capacity (TAC), mmol/L | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Assessed using the ABTS+ radical cation decolorization assay with spectrophotometric analysis.
Ferric Reducing Ability of Plasma (FRAP), mmol/L | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Quantified using the FRAP assay, based on the reduction of Fe3+ to Fe2+, measured at 593 nm.
Heat Shock Protein 70 (HSP70), ng/mL | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Plasma concentrations will be measured using sandwich-type enzyme-linked immunosorbent assay (ELISA), with detection at 450 nm after chromogenic substrate reaction.
Fibronectin, µg/mL | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Quantified by high-sensitivity ELISA using monoclonal antibodies specific for fibronectin. Detection will be performed at 450 nm, using manufacturer-calibrated standard curves.
Laminin, µg/mL | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Determined by validated ELISA sandwich assay with photometric quantification at 450 nm. Assay will be conducted in duplicate with quality controls and external calibrators.
Plasma Ceramides, ng/mL | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Quantified using liquid chromatography-tandem mass spectrometry (LC-MS/MS) after lipid extraction via the Folch method. Identification and quantification will be based on retention times and certified external standards.
Plasma Sphingolipids, ng/mL | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Plasma concentrations will be determined using validated LC-MS/MS protocols with external calibrators, after sample preparation by chloroform/methanol extraction.
Plasma Cardiolipins, ng/mL | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Quantified by LC-MS/MS using C18 chromatographic separation and tandem MS detection, with identification based on spectral patterns and standard curves.
Plasma Prostaglandins, pg/mL | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Determined by LC-MS/MS with high-sensitivity detection and external calibration for absolute quantification. Sample preparation follows established lipidomic protocols.
Plasma Leukotrienes, pg/mL | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  Measured using targeted LC-MS/MS following Folch lipid extraction. Identification and quantification will be conducted against authentic leukotriene standards.
Pancreatic Remnant Volume, cm³ | Day 0 (preoperative), 3 months post-discharge, 6 months post-discharge
  The remnant pancreatic volume will be measured using computed tomography (CT) and/or magnetic resonance imaging (MRI). Volumetric analysis will be performed through three-dimensional segmentation using 3D Slicer software.

CONTACTS AND LOCATIONS:
Overall Officials: Marco A Ribeiro, PhD, MSc, BSc, RD, Principal Investigator — Ribeirão Preto Medical School University of São Paulo; Anderson M Navarro, Prof, PhD, MSc, BSc, RD, Study Director — Ribeirão Preto Medical School University of São Paulo
Locations (1):
- Ribeirão Preto Medical School University of São Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to ethical considerations and institutional policy regarding data confidentiality. The dataset contains sensitive health information, and there are no current plans or infrastructure in place for secure external sharing.

REFERENCES:
- See also: Official website of the Ethics Committee - Hospital das Clínicas, Ribeirão Preto Medical School (HCRP-USP). — https://site.hcrp.usp.br/comite-de-etica/
- See also: Official website of the Ribeirão Preto Medical School, University of São Paulo (FMRP-USP). — https://www.fmrp.usp.br/en/